CLINICAL TRIAL: NCT03191656
Title: A Post-Market Clinical Follow-up Study to Evaluate the Corvia Medical, Inc. InterAtrial Shunt Device - IASD® System II to REDUCE Elevated Left Atrial Pressure in Patients With Heart Failure
Brief Title: REDUCE LAP-HF III Corvia Protocol 1701
Acronym: REDUCELAPHFIII
Status: Recruiting | Type: Observational
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1701
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: IASD Implant — Implantation of the IASD device using trans-septal puncture and the IASD system

SUMMARY:
This is a post market trial to be conducted at sites in Germany. The device has CE approval in the EU. The purpose of this observational registry is to collect post market data in consecutive patients treated with the IASD System II, to further evaluate efficacy, safety and quality of life outcomes as a new treatment for patients with heart failure in a "real world" practice setting.

ELIGIBILITY:
This is a post market registry so no criteria requirements (only recommendations).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with preserved (HFpEF) or mid-range ejection fraction (HFmrEF) with elevated left atrial pressures, who remain symptomatic despite standard Guideline Directed Medical Therapy (GDMT), in accordance with CE-mark approved labeling.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 days
  Device and or procedure related serious adverse cardiac events
New York Heart Classification | 12 months
  Improvement in NYHA Classification
Quality of Life Improvement (KCCQ score) | 12 months
  Improvement in KCCQ score
Quality of Life Improvement (EQ5D) | 12 months
  Improvement in EQ5D score

CONTACTS AND LOCATIONS:
Locations (27):
- Germany (26):
  - Herzzentrum der Kerckhoff-Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen Klinik für Kardiologie, Bad Oeynhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Unfallkrankenhaus Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Herzzentrum der Universität zu Köln, Cologne
  - Klinikum Lippe GmbH, Detmold
  - Herzzentrum Dresden GmbH, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Kardiologie, Pneumologie u. Angiologie, Düsseldorf
  - Elisabeth-Krankenhaus Essen, Essen
  - Universitätsklinikum Gießen, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Universitäts Klinikum Halle, Halle
  - Klinikum am Plattenwald Bad Friedrichshall, Heilbronn
  - Klinikum Karlsburg, Karlsburg
  - Klinik für Innere Medizin III mit den Schwerpunkten Kardiologie, Angiologie und internistische, Kiel
  - Klinikum Sankt Georg, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Munster, Münster
  - Niels-Stensen-Kliniken - Marienhospital, Osnabrück
  - St Vincenz-Kranenhaus, Paderborn
  - Herz-Kreislauf-Zentrum Rotenburg, Rotenburg (Wümme)
  - Helios Kliniken Schwerin, Schwerin
  - Universitätsklinik Ulm-Keßler, Ülm
  - Evangelisches Krankenhaus Paul Gerhardt Stift - Unfallstation, Wittenberg
  - Heinrich Braun Klinikum, Zwickaü
- Bürgelspital Solothurn, Solothurn, Switzerland